CLINICAL TRIAL: NCT01078922
Title: A Phase II Open-label Study of Single Agent Ofatumumab in Patients With Relapsed and/or Refractory Diffuse Large B Cell Non Hodgkin Lymphomas
Brief Title: Patients With Relapsed or Refractory Diffuse Large B Cell Non Hodgkin Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow acrual
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OFT113588 (0908)
Record Dates: First submitted 2010-02-23; First posted 2010-03-02 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Non-Hodgkin Lymphomas
Keywords: ofatumumab diffuse B cell non hodgkins lymphoma DLBCL; refractory DLBCL; relapsed DLBCL
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): The first dose administered of ofatumumab should be 300 mg to minimize infusion reactions. The initial rate of the first infusion of 1000 mg ofatumumab (0.3mg/ml) should be 12ml/h. If no infusion reactions occur the infusion rate should be increased every 30 minutes, to a maximum of 400 ml/h. If this schedule is followed, the infusion duration will be approximately 4.5 hours.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — The first dose administered of ofatumumab should be 300 mg to minimize infusion reactions. The initial rate of the first infusion of 1000 mg ofatumumab (0.3mg/ml) should be 12ml/h. If no infusion reactions occur the infusion rate should be increased every 30 minutes, to a maximum of 400 ml/h. If this schedule is followed, the infusion duration will be approximately 4.5 hours.
  Other Names: OFT113588

SUMMARY:
This is a phase II open label study that looks at the efficacy and toxicity of Ofatumumab monotherapy in patients with relapsed and/or refractory diffuse large B-cell lymphoma (DLBCL). Patients will receive weekly infusions of Ofatumumab of 1000 mg each for 8 weeks (induction phase) followed by continuing the study drugs every other week in subsequent cycles (maintenance phase). Each 4 weeks of therapy will be calculated as one cycle. Treatment will continue until disease progression, toxicity, patient's withdrawal, or investigator's discretion.

DETAILED DESCRIPTION:
Ofatumumab is a fully human monoclonal IgG1κ-antibody targeting a novel cluster of differentiation antigen 20(CD20)-epitope. Preclinical data show that ofatumumab is active against B-cell lymphoma/chronic lymphocytic leukemia cell-lines with low CD20-antigen density and an increased expression of complement inhibitory molecules. Ofatumumab was superior to rituximab in its ability to induce lysis in B-cell lines and also killed fresh B-chronic lymphocytic leukemia cells that were resistant to rituximab. Ofatumumab has a slower off-rate and more stable CD20 binding in comparison with rituximab and targets a different epitope of the CD20 antigen than rituximab [Teeling, 2004, Teeling, 2006]. In cynomolgus monkeys, the duration of B-cell depletion from peripheral blood and lymph nodes induced by ofatumumab was longer than that of rituximab [Dechant, 2003].

Ofatumumab's ability to induce complement-dependent cytotoxicity (CDC) has been specifically studied in isolated lymphoma cells from chemotherapy refractory DLBCL patients [Cillessen, 2007]. Ofatumumab and rituximab induced CDC of all DLBCL samples tested, including the DLBCL cell lines SUDHL-4, SUDHL-5 and HT and lymphoma cells derived from ten chemotherapy-refractory DLBCL patients.

Ofatumumab was significantly more effective in inducing CDC in nine of the ten DLBCL tumor samples when compared with rituximab (p=0.001). The lethal doses (LD50) for ofatumumab (0.1 ± 2.8 μg/mL) were significantly lower when compared with the LD50 for rituximab (6.4 ± 4.9μg/mL, p=0.04). Sensitivity of DLBCL patient cells to ofatumumab- and rituximab-induced CDC negatively correlated with expression of complement defense molecule CD59, but not with expression of CD46 or CD55. Functional inhibition of CD55 and CD59 using blocking mAb demonstrated that ofatumumab-induced CDC of DLBCL tumor cells was less sensitive to expression of these complement defense molecules than rituximab-induced CDC.

Thus, chemotherapy-refractory DLBCL cases are sensitive to CD20 mAb-induced CDC with ofatumumab being the most effective mAb, especially in patients expressing high levels of CD59.

Safety and efficacy of ofatumumab, has been analyzed in multicenter dose-escalating phase I/II studies in chronic lymphocytic leukemia (CLL) and follicular lymphoma (FL). Three cohorts of patients including 33 patients with relapsed or refractory CLL received weekly infusions of ofatumumab for four weeks as follows: cohort A, the first infusion was 100 mg and three subsequent infusions of 500 mg; cohort B, the first infusion was 300 mg and three subsequent infusions of 1000 mg; cohort C, the first infusion was 500 mg and three subsequent infusions of 2000 mg. The maximum tolerated dose was not reached. The majority of related adverse events occurred at first infusion, and the number of adverse events decreased at each subsequent infusion. Seventeen (51%) of 33 patients experienced infections, 88% of them of grade 1-2. One event of interstitial pneumonia was fatal; all other cases resolved within one month. The response rate in cohort C was 50% (13/26 patients) [Coiffier, 2008].

Interim data from a single arm study in refractory CLL was presented at ASH 2008 [Osterborg, 2008]. The activity of ofatumumab was evaluated in 138 patients with refractory CLL: 59 were refractory to both fludarabine and alemtuzumab (double-refractory: DR) and 79 were refractory to fludarabine and considered inappropriate candidates for alemtuzumab due to bulky tumor in their lymph nodes (bulky fludarabine-refractory: BFR group). Patients received 8 weekly infusions of ofatumumab followed by 4 monthly infusions. The first dose was 300mg, doses 2-12 were 2000 mg. Median time to next CLL therapy was 9 months for the DR group and 8 months for the BFR group. The median overall survival was about 14 months for the DR group and 15 months for the BFR group. Response at week 12 was significantly correlated with longer survival for both groups. Ofatumumab was associated with infusion-related adverse events on the first infusion day in 46% of patients in the DR group and 38% in the BFR group, which were grade 3 in 7% and 3% of events, respectively. There were no grade 4 infusion-related events. These events generally subsided with subsequent infusions.

The most common grade 3 or 4 toxicities were infections (25% in DR; 27% in BFR group) and hematologic events including neutropenia (12% in DR; 10% in BFR group) and anemia (8% in DR; 4% in BFR group). Death within 8 weeks from start of treatment occurred in 2 patients (3%) in the DR group (sepsis, n=1; fungal pneumonia, n=1) and 3 patients (4%) in the BFR group (PD, n=1; sepsis, n=1; myocardial infarction, n=1).

In a phase I/II study evaluating safety and efficacy of ofatumumab in relapsed or refractory FL grade 1-2, 4 dose-groups of 10 patients received 4 weekly infusions of 300, 500, 700, or 1000 mg [Hagenbeek, 2008]. Patients had a median of two prior FL therapies and 13% had elevated lactate dehydrogenase (LDH). No safety concerns or maximum tolerated dose were identified. Most adverse events occurred on the first infusion day and were common toxicity criteria (CTC) grade 1-2. Eight related events were grade 3. Treatment caused immediate and profound B-cell depletion. The response rate was not dose dependent (dose expressed as mg/patient, mg/kg body weight or body surface area (mg/m2)) with responses obtained in all 4 dose groups (300 mg: 5 of 8 subjects (63%); 500 mg: 3 of 10 subjects (30%); 700 mg: 2 of 10 subjects (20%); and 1000 mg: 5 of 10 subjects (50%). Median time to progression (TTP) for all patients was 8.8 months. Median TTP for responders, duration of response, and time to next anti-FL therapy has not been reached at a median follow-up of 9.2 months. Ofatumumab was able to induce responses in 8 of 14 patients relapsing following rituximab, including 3 of 4 rituximab refractory patients.

Ofatumumab is currently being evaluated in patients with rituximab-refractory FL (Hx-CD20-405), relapsed DLBCL (GEN-415), rituximab-relapsed/refractory DLBCL in combination with salvage chemotherapy (OMB110927) and in a phase III trial in relapsed/refractory DLBCL (OMB110928) at a dose of 1000mg, and in combination with chemotherapy in FL (Hx-CD20-409) at doses of 500mg and 1000mg.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and/or refractory DLBCL,not HSCT candidates. Pts must have failed standard of care (SOC) therapy w/rituximab plus CHOP or its equivalent & not considered hematopoietic stem cell transplant (HSCT) candidates based on investigator's discretion
* Pts must have measurable disease radiographically on CT and/or PET scans and/or bone marrow biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Age ≥18 years. No upper limit of age
* Life expectancy of 6 months or more based on investigator's best estimate.
* Pts able to read, understand, & sign informed consent
* Evidence of CD20 positivity in treated pts, using flow or immunohistochemistry.
* Pts will be stratified based on bulk of disease (bulk defined as any area w/ more than 5cm in greatest dimension)
* Pts must agree to an acceptable form of birth control

Exclusion Criteria:

* Other histologies of non-Hodgkin's lymphoma (NHL)
* Known central nervous system (CNS) involvement with NHL
* Known HIV positive status
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment.
* Corticosteroid use is allowed as long as it is for non-lymphoma related causes such as rheumatoid arthritis and chronic obstructive pulmonary disease (COPD).
* Pts w/prior malignancies are allowed as long as they are in remission & their last treatment for such malignancy is 2 years prior to enrollment or more. Pts w/non-melanoma skin cancers that have received adequate therapy prior to enrollment & women w/history of cervical cancers are allowed.
* Significant concurrent uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurologic, cerebral, or psychiatric disease.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per the investigator's assessment).
* Adequate bone marrow function by virtue of having Platelets >50,000/ul & absolute neutrophil count (ANC) >1000/ul is required unless low counts are attributed to diffuse bone marrow infiltration with NHL as documented with a bone marrow biopsy exam.
* Pts with creatinine >2.0 times the upper limit of normal will be excluded unless they have a normal creatinine clearance-estimated or measure 12 or 24 hour creatinine clearance of <60 mL/min
* Pts w/total bilirubin >1.5 times upper limit of normal will be excluded, unless due to DLBCL involvement of liver or a known history of Gilbert's disease.
* Pts with aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/Alkaline phosphatase (Alk Phos) >2.5 times upper limit of normal
* Previous tx with Ofatumumab
* Prior exposure to an investigational agent within 4-weeks from starting Ofatumumab
* History of significant cerebrovascular disease or event w/significant symptoms or sequelae
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to randomization, congestive heart failure (NYHA III-IV), & arrhythmia unless controlled by therapy, w/exception of extra systoles or minor conduction abnormalities.
* Positive serology for hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive & regardless of HBsAb status, a HB DNA test will be performed and if positive the subject to be excluded. Note: If HBcAb positive and HBsAb positive, which is indicative of a past infection, subject can be included
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result.
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening, including women whose last menstrual period was less than 1 year prior to screening, unable or unwilling to use adequate contraception from study start to 1 year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, S.C.
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Oncology Specialists, S.C, Niles, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ofatumumab
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR)
Description: OR = # of patients with a Complete Response (CR) plus # of patients with a Partial Response (PR) divided by the total # of evaluable patients.
  A CR is defined as:
  1. Disappearance of all disease.
  2. If nodal masses that Positron Emission Tomography (PET)- positive prior to therapy; they must be PET negative
  3. If the nodal masses were Variably or PET negative; they must regress to normal.
  4. No palpable liver or spleen
  5. Palpable nodal masses are no longer palpable
  6. Negative bone marrow biopsy
  A PR is defined as:
  1. Regression of measurable disease and no new sites of disease.
  2. > 50% decrease in Sum of Product of Diameters (SPD) of up to 6 largest masses with no increase in the size of other nodes. If the nodal masses were PET positive prior to therapy then PET positive at previously involved sites is allowed. If they were Variably or PET negative then regression on CT is required.
  3. No increase in the size of the liver or spleen
Time Frame: evaluated every 2 months up to 80 weeks
Population: Analysis was per protocol. Patients were evaluated every 2 cycles for Overall Response, up to 80 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 11
percentage of participants | 18

2. Secondary Outcome: Overall Clinical Benefit (OCB)
Description: OCB = # patients with a CR + # of patients with a PR + # patients with Stable Disease (SD) divided by the number of evaluable patients CR and PR is defined in Outcome Measure #1
  SD is defined as:
  1. Failure to attain CR/PR or Progressive Disease (PD)
  2. PET remains positive.
  PD is defined as:
  1. Any new lesion > 1.5 cm in longest axis
  2. An increase 50% or more of previously involved sites from nadir
  3. 50% increase in SPD of more than one node or 50% increase in the longest diameter of a previously identified node that is > 1 cm in shortest axis
  4. PET remains positive if it was positive before therapy.
Time Frame: Evaluated every 2 cycles (every 2 months), up to 80 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 11
percentage of participants | 36

ADVERSE EVENTS:
Arm/Group | Ofatumumab
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=11)
Pain (General disorders) | 1
Graft versus host disease (General disorders) | 1 (2)
Vertigo (General disorders) | 1
Subcapsular liver hemorrhage (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Reflux esophagitis (Gastrointestinal disorders) | 1
Death-disease progression (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=11)
Alkaline Phosphatase (Blood and lymphatic system disorders) | 2
anemia (Blood and lymphatic system disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 6
Anxiety (Psychiatric disorders) | 1
Alopecia (General disorders) | 4
Abdominal discomfort (General disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
increased bilirubin (Renal and urinary disorders) | 1
bacteremia (Infections and infestations) | 1
increased creatinine (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 2
Chills (General disorders) | 2
cold (Infections and infestations) | 2
conjunctival irritation (Eye disorders) | 1
cramps (Musculoskeletal and connective tissue disorders) | 1
depression (Psychiatric disorders) | 1
diarrhea (Gastrointestinal disorders) | 5
dry mucous membranes (General disorders) | 2
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 1
edema (Vascular disorders) | 4
epigastric pain (Gastrointestinal disorders) | 1
eye pain (Eye disorders) | 1
eye edema (Eye disorders) | 1
fatigue (General disorders) | 6
fever (Infections and infestations) | 2
flushing to face (General disorders) | 1
gastritis (Gastrointestinal disorders) | 1
hemorroids (Gastrointestinal disorders) | 1
headache (Nervous system disorders) | 1
increased heart rate (Cardiac disorders) | 1
hypocalcemia (Blood and lymphatic system disorders) | 3
hypokalemia (Blood and lymphatic system disorders) | 3
hyponatremia (Blood and lymphatic system disorders) | 4
hypoalbuminemia (Gastrointestinal disorders) | 3
hypomagnesemia (Blood and lymphatic system disorders) | 1
hyperglycemia (Endocrine disorders) | 2
hyperkalemia (Blood and lymphatic system disorders) | 1
hypertension (Cardiac disorders) | 2
hypercalcemia (Blood and lymphatic system disorders) | 1
insomnia (General disorders) | 2
itchiness (Skin and subcutaneous tissue disorders) | 2
infection (Infections and infestations) | 1
leukopenia (Blood and lymphatic system disorders) | 3
lyphmopenia (Blood and lymphatic system disorders) | 4
neck stiffness (Musculoskeletal and connective tissue disorders) | 1
nervousness (Psychiatric disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 4
nasal congestion (General disorders) | 1
neuropathy (Nervous system disorders) | 4
nausea (Gastrointestinal disorders) | 5
night sweats (General disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
pain (General disorders) | 6
parasthasia lower extremities (General disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 2
sinus pressure (General disorders) | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
skin tears (Skin and subcutaneous tissue disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 2
taste alteration (Gastrointestinal disorders) | 1
throat scratchy (Gastrointestinal disorders) | 1
urinary tract infection (Infections and infestations) | 1
ulcer (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 5
viral infection (Gastrointestinal disorders) | 1
vocal cord paralysis (General disorders) | 1
watery eyes (Eye disorders) | 1
weakness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No